CLINICAL TRIAL: NCT07357376
Title: Evaluating a Non-Opioid Analgesic Strategy for Enhanced Recovery After Total Knee Arthroplasty: A Randomized Controlled Trial of Suzetrigine
Brief Title: Evaluating Suzetrigine for Pain Control Following TKA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: American Association of Hip and Knee Surgeons (Other)
Responsible Party: Principal Investigator, Teja Yeramosu, Resident Physician, AdventHealth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-ORTHO-JOURNAVX-01
Record Dates: First submitted 2026-01-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Following Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Postoperative Pain; Journavx; Suzetrigine; Opioid; Enhanced Recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suzetrigine/Journavx (Experimental)
  Interventions: Drug: Suzetrigine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suzetrigine — Suzetrigine is an oral, non-opioid pain medication that works by blocking specific sodium channels involved in pain signaling. In this study, participants assigned to the suzetrigine group will receive a 100 milligram oral dose in the preoperative area, immediately prior to undergoing the procedure, followed by 50 milligrams taken by mouth twice daily for 14 days after surgery. Suzetrigine will be given in addition to standard postoperative pain care, including acetaminophen, nonsteroidal anti-inflammatory drugs when appropriate, and opioid pain medication only if needed for breakthrough pain.
  Arms: Suzetrigine/Journavx
Drug: Placebo — The placebo is an oral tablet designed to look like the suzetrigine tablet but contains no active drug. In this study, participants assigned to the placebo group will receive a tablet in the preoperative area immediately prior to the procedure, followed by placebo tablets taken by mouth twice daily for 14 days after surgery. The placebo will be given in addition to standard postoperative pain care, including acetaminophen, nonsteroidal anti-inflammatory drugs when appropriate, and opioid pain medication only if needed for breakthrough pain.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if a non-opioid pain medicine called suzetrigine works to treat pain after total knee replacement surgery in adults. It will also learn about the safety of suzetrigine. The main questions it aims to answer are:

Does suzetrigine lower the amount of opioid pain medicine participants use after surgery?

Does suzetrigine have any effect on postoperative patient-reported outcomes, including pain scores, range of motion, length of stay, and KOOS/PROMIS surveys?

Researchers will compare suzetrigine to a placebo to see if suzetrigine works to treat pain after total knee replacement surgery.

Participants will:

Take suzetrigine or a placebo by mouth for 14 days after surgery

Receive standard pain care, including opioid pain medicine only if needed

Report their pain levels using short daily surveys

Attend routine follow-up visits after surgery

DETAILED DESCRIPTION:
Post-operative pain management following total knee arthroplasty (TKA) continues to present significant challenges. Despite multimodal Enhanced Recovery After Surgery (ERAS) protocols, over 60% of patients still require opioid medications two weeks after surgery. Given the ongoing opioid epidemic, opioid prescribing is a priority for quality improvement in orthopaedic surgery. High opioid exposure is associated with constipation, nausea, increased risk of falls, hindered rehabilitation, and persistent opioid use. Furthermore, opioid use within the early postoperative period following TKA is associated with a dose-dependent increased risk of periprosthetic joint infection and venous thromboembolic events. With over 700,000 TKAs performed each year in the United States, these complications represent not only individual patient risks but also broader public health concerns.

Multimodal pain regimens consisting of alternative analgesics such as acetaminophen, NSAIDs, and gabapentinoids may only provide partial relief for patients, leaving opioids as the default choice for managing breakthrough pain, despite their undesirable side effect profile and addictive potential.[8] This ongoing challenge underscores the urgent need to identify safer and more effective pain management strategies.

Suzetrigine (Brand name: Journavx), a selective inhibitor of NaV1.7/NaV1.8 channels, has emerged as a promising candidate. Phase 3 clinical trials have shown that suzetrigine provides pain relief comparable to opioids, effectively reducing pain scores, with fewer adverse effects. Data from phase 2 bunionectomy studies further support its opioid-sparing capabilities. Unlike opioids, suzetrigine does not cause sedation, respiratory depression, or dependency. Its favorable pharmacokinetic properties, including renal-sparing metabolism and convenient oral twice-daily dosing, make it well-suited for integration into ERAS protocols.

The purpose of this randomized controlled trial is to assess whether suzetrigine can serve as an effective, opioid-sparing analgesic after TKA. If the results are successful, this could lead to expanded FDA labeling, wider adoption in orthopaedic practices, and a significant decrease in opioid prescriptions on a large scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for elective, unilateral primary total knee arthroplasty
* Able to tolerate oral medications after surgery

Exclusion Criteria:

* Revision or bilateral total knee arthroplasty
* American Society of Anesthesiologists (ASA) physical status classification greater than 3
* Severe renal impairment (estimated glomerular filtration rate less than 15 mL/min/1.73 m²)
* Severe hepatic impairment (Child-Pugh Class C)
* Chronic opioid use of 30 morphine milligram equivalents per day or greater for more than 3 months
* Pregnancy or breastfeeding
* Seizure disorder or known hypersensitivity to suzetrigine
* Use of medications contraindicated with CYP3A metabolism
* Active gastrointestinal ulcer or bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Usage | 2 weeks
  MME of opioid usage

SECONDARY OUTCOMES:
Numeric Pain Rating Scale Scores | 2 Weeks
  Pain will be measured using the Numeric Pain Rating Scale (NPRS), a patient-reported pain scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate worse pain. NPRS scores will be collected daily for the first 14 days after surgery and summarized over the 2-week postoperative period.
Range of Motion | 2 Weeks
  Knee range of motion will be assessed using goniometric measurement of knee flexion, performed by a trained care provider during routine postoperative evaluations. Range of motion reflects the degree of knee movement achieved after surgery. Greater range of motion indicates better functional recovery. Measurements will be obtained at discharge and at the 2-week postoperative visit.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score | 2 Weeks
  Pain-related interference with daily activities will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference questionnaire. This is a standardized patient-reported outcome measure that evaluates the extent to which pain interferes with physical, social, and emotional functioning. Higher scores indicate worse pain interference.
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Score | 2 Weeks
  Physical function will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function questionnaire, a validated patient-reported measure of mobility and functional ability. Higher scores indicate better physical function.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 Weeks
  Knee-related symptoms and function will be assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire. This patient-reported outcome measure evaluates pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Higher scores indicate better knee-related outcomes.
Incidence of Treatment-Emergent Side Effects | 2 Weeks
  The occurrence of treatment-emergent side effects will be assessed during the first 2 weeks after surgery. Side effects monitored include nausea, vomiting, constipation, dizziness, sedation, pruritus, headache, weakness, and worsened sleep. The outcome will be reported as the number of participants experiencing one or more side effects during the assessment period. A higher number of participants with side effects indicates worse tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Ramakanth Yakkanti, MD, Principal Investigator — Rothman Orthopaedics Florida at AdventHealth

IPD SHARING:
Plan to Share IPD: No
Individual participant data may not be shared outside the research team. The study includes sensitive health information collected under institutional review board approval, and participant consent does not include public data sharing. Data will be analyzed and reported in aggregate to protect participant privacy.

REFERENCES:
- [Background] Hu S, Lyu D, Gao J. Suzetrigine: The first Nav1.8 inhibitor approved for the treatment of moderate to severe acute pain. Drug Discov Ther. 2025 Mar 6;19(1):80-82. doi: 10.5582/ddt.2025.01010. Epub 2025 Feb 27. PMID 40010720
- [Background] Hang Kong AY, Tan HS, Habib AS. VX-548 in the treatment of acute pain. Pain Manag. 2024 Sep;14(9):477-486. doi: 10.1080/17581869.2024.2421749. Epub 2024 Nov 18. PMID 39552600
- [Background] Hannon CP, Fillingham YA, Nam D, Courtney PM, Curtin BM, Vigdorchik JM, Buvanendran A, Hamilton WG, Della Valle CJ; AAHKS Anesthesia & Analgesia Clinical Practice Guideline Workgroup. Opioids in Total Joint Arthroplasty: The Clinical Practice Guidelines of the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. J Arthroplasty. 2020 Oct;35(10):2709-2714. doi: 10.1016/j.arth.2020.05.034. Epub 2020 May 26. No abstract available. PMID 32571594
- [Background] Shichman I, Roof M, Askew N, Nherera L, Rozell JC, Seyler TM, Schwarzkopf R. Projections and Epidemiology of Primary Hip and Knee Arthroplasty in Medicare Patients to 2040-2060. JB JS Open Access. 2023 Feb 28;8(1):e22.00112. doi: 10.2106/JBJS.OA.22.00112. eCollection 2023 Jan-Mar. PMID 36864906
- [Background] Chung BC, Bouz GJ, Mayfield CK, Nakata H, Christ AB, Oakes DA, Lieberman JR, Heckmann ND. Dose-Dependent Early Postoperative Opioid Use Is Associated with Periprosthetic Joint Infection and Other Complications in Primary TJA. J Bone Joint Surg Am. 2021 Aug 18;103(16):1531-1542. doi: 10.2106/JBJS.21.00045. PMID 34043598
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Sabatino MJ, Kunkel ST, Ramkumar DB, Keeney BJ, Jevsevar DS. Excess Opioid Medication and Variation in Prescribing Patterns Following Common Orthopaedic Procedures. J Bone Joint Surg Am. 2018 Feb 7;100(3):180-188. doi: 10.2106/JBJS.17.00672. PMID 29406338
- [Background] Atwood K, Shackleford T, Lemons W, Eicher JL, Lindsey BA, Klein AE. Postdischarge Opioid Use after Total Hip and Total Knee Arthroplasty. Arthroplast Today. 2021 Jan 30;7:126-129. doi: 10.1016/j.artd.2020.12.021. eCollection 2021 Feb. PMID 33553537
- [Background] Dawson Z, Stanton SS, Roy S, Farjo R, Aslesen HA, Hallstrom BR, Bicket MC. Opioid Consumption After Discharge From Total Knee and Hip Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2024 Aug;39(8):2130-2136.e7. doi: 10.1016/j.arth.2024.01.063. Epub 2024 Feb 8. PMID 38336301
- [Background] Shah R, Kuo YF, Westra J, Lin YL, Raji MA. Opioid Use and Pain Control After Total Hip and Knee Arthroplasty in the US, 2014 to 2017. JAMA Netw Open. 2020 Jul 1;3(7):e2011972. doi: 10.1001/jamanetworkopen.2020.11972. No abstract available. PMID 32729917